CLINICAL TRIAL: NCT06849739
Title: Study on the Correlation and Consistency of Measuring Biologic Drug Plasma Concentrations Based on Different Detection Methods
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-563
Record Dates: First submitted 2024-11-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- infliximab group: IBD patients using infliximab
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)
- adalimumab group: IBD patients using adalimumab
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)
- vedolizumab group: IBD patients using vedolizumab
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)
- ustekinumab group: IBD patients using ustekinumab
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)

INTERVENTIONS:
Drug: biologic therapy(eg:IFX,ADA,UST,VDZ) — This study compares the detection of blood samples from IBD patients after biologic therapy(eg:IFX,ADA,UST,VDZ) using different methods

SUMMARY:
In recent years, biologics (such as infliximab, adalimumab, vedolizumab, and ustekinumab) have shown great potential in the treatment of inflammatory bowel disease (IBD), transforming the traditional treatment model for IBD. Despite achieving good efficacy, some patients do not respond to biologics, which may be related to low drug concentrations in the blood. Guidelines recommend therapeutic drug monitoring (TDM) during the treatment of IBD. Currently, many commercial testing methods are available to detect the trough levels of biologics; however, data on the diagnostic accuracy and practicality of these methods remain limited. This study compares the detection of blood samples from IBD patients after administration using ELISA, PICA, and CLIA methods, aiming to provide more accurate guidance and evidence for TDM in Chinese IBD patients undergoing biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older; diagnosed with inflammatory bowel disease according to the 2019 European ECCO-ESGAR guidelines; who have not previously received any biologic therapy or, based on the treating physician's judgment, require treatment with infliximab (IFX), adalimumab (ADA), vedolizumab (VDZ), or ustekinumab (UST) .

Exclusion Criteria:

* Patients who refuse treatment with infliximab, adalimumab, vedolizumab, or ustekinumab for various reasons, or those with contraindications; patients currently using antibiotics or who have been in contact with probiotics/antibiotics in the past month; those with concomitant active autoimmune diseases, active tumors, etc.; those with severe oral diseases; patients experiencing other diseases unrelated to inflammatory bowel disease during treatment but may affect the efficacy of inflammatory bowel disease treatment; pregnant or lactating women; those deemed unsuitable for participation in this study by the investigator's judgment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Based on the treating physician's judgment, IBD patients require biologic therapy with infliximab (IFX), adalimumab (ADA), vedolizumab (VDZ), or ustekinumab (UST) .
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
plasma concentration | During hospitalization for biologic injections，an average of 1 week
  plasma concentration refers to the total concentration of a biologic drug（such as infliximab, adalimumab, vedolizumab, and ustekinumab） in the plasma after absorption.

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided